CLINICAL TRIAL: NCT03782337
Title: The Predictors and Benefits of Multi-discipline Disease Management Program in Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8H1271
Record Dates: First submitted 2018-12-05; First posted 2018-12-20 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure With Decompensation
Keywords: Heart failure,; Cardiac biomarker; Cardiopulmonary exercise test; Multi-discipline disease management program; Reverse remodeling
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Biomarkers for cardiovascular disease, e.g., sST2, GDF15, and DNA testing for arrhythmogenic cardiomyopathy.
  2. Cytokines, e.g., inflammation cytokines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: multi-discipline disease management program — The multi-discipline disease management program consists of nursing lead education program, dietitian consultation, psychologist consultation and assessment, and cardiac rehabilitation program by physical therapist.The cardiovascular lead nurse will contact the patient by telephone within 3 days after discharge. An appointment at the outpatient clinic will be arranged within 1 to 2 weeks after discharge. The purposes of the telephone call are to reinforce self-management and recognition of HF symptoms and to screen post-discharge health status.

SUMMARY:
The investigator will investigate the predictors includes cardiac biomarkers, endothelial function and cardiopulmonary exercise test in prediction of cardiovascular outcome in patients with heart failure discharged from hospital.

DETAILED DESCRIPTION:
Background: Readmission and mortality are high after heart failure (HF) hospitalization. Heart Failure Multi-discipline disease management program (HFDMP) has shown to decrease 30% in readmission for decompensated heart failure or other cardiovascular causes. This was associated with a decreased in medical cost of care and a trend towards a lower mortality rate. Despite evidence that HFDMPs is effective, however, they are not widely employed in Taiwan. Some HFDMPs did not show improved health status compared with usual care. The "best way" to design and implement a HFDMP is not clear. It is still not clear if HFDMP would benefit all heart failure patients or should instead be targeted to specific subsets. Lysyl oxidase-like 2 (Loxl2) is enzyme, which crosslinks collagen in fibrotic processes such like liver cirrhosis or lung fibrosis. Recently, Lysyl oxidase-like 2 (Loxl2) was also found to participate the process of cardiac interstitial fibrosis and heart failure. Interestingly, the serum level of Loxl2 is in good correlation with the severity of heart failure. However, there is still unknown whether Loxl2 is useful biomarker for predicting the long-term outcome in patient with heart failure. From the mechanism of Loxl2 in the process of heart failure, the serum level of Loxl2 may be a good maker for predict the degree of cardiac remodeling. Our animal study showed the correlation between myocardial fibrosis and Loxl2 serum level. Therefore, The investigator will investigate whether serum Loxl2 level is a good maker for predictor the long-term outcome in patient with heart failure and predictor of cardiac remodeling. The correlation between this novel cardiac biomarker and endothelial function, cardiopulmonary function test will also be evaluated.

Objectives: The investigator will investigate the predictors includes cardiac biomarkers ( such as serum Loxl2 level, B-type natriuretic peptide (BNP), soluble ST2), endothelial function and cardiopulmonary exercise test in prediction of cardiovascular outcome and reverse remodeling in patients with heart failure discharged from hospital.

Design: A prospective cohort study

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent before any assessment is performed.
2. Inpatients ≥ 18 years of age, male or female.
3. Patients with a diagnosis of heart failure New York Heart Association (NYHA) class II-IV with BNP >100 pg/mL

Exclusion Criteria:

1. Estimated survival time < 6 months
2. Long-term bedridden more than 3 months
3. Cannot tolerance exercise test due to muscular skeletal disorder
4. Cannot co-operate all functional studies
5. Ventilator dependent
6. Terminal heart status
7. Family reject to participate this project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients population who admitted to a referred medical center.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants That Had First Occurrence of the Composite Endpoint, Which is Defined as Either Cardiovascular (CV) Death or Heart Failure (HF) Readmission | up to 36 months
  Number of participants that had first occurrence of the composite endpoint, which is defined as either CV death or HF readmission.

SECONDARY OUTCOMES:
Change From Baseline to Month 6 and Month 12 for the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ 12) Clinical Summary Score | Baseline, Month 6 , Month 12
  Change from baseline to Month 6 and month 12 for the Kansas City Cardiomyopathy Questionnaire short form (KCCQ12) clinical summary score. KCCQ12 is a 12-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ12 clinical summary score is a composite assessment of physical limitations and total symptom scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Number of Participants - All-cause Mortality | up to 36 months
  Number of patients - All-cause mortality. All-cause mortality is common in Heart Failure (HF) patients. This measures how many patients had this event.
Number of Participants with changes in ventricular shape using echocardiographic endocardial surface analysis techniques | 12 months
  Number of Participants with changes in ventricular shape using echocardiographic endocardial surface analysis techniques from patient discharge to 12 months after

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Ming Chen, MD, Principal Investigator — Chang Gung Memorial Hospital Heart Failure Center
Locations (1):
- Chang Gung Memorial Hospital Heart Failure Center, Kaohsiung City, Bird Pine Area, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss with other investigators about individual participant data (IPD) sharing.